CLINICAL TRIAL: NCT04640051
Title: Preprocedural Assessment of Anatomy and Device Sizing With CT and 3D Simulation in Left Atrial Appendage Occlusion: the PRECISE LAAO Registry
Brief Title: Preprocedural Assessment of Anatomy and Device Sizing With CT and 3D Simulation in Left Atrial Appendage Occlusion.
Acronym: PRECISE LAAO
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Ian Buysschaert, MD PhD, Principal Investigator, AZ Sint-Jan AV
Other Study IDs: version 1.0 26/10/2020
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: LAAO With Amplatzer Amulet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAAO group: Patients scheduled for LAAO with Amplatzer Amulet (Abbott) and for whom a 3D in silico simulation by FEops HEARTguide is available and reviewed before implantation
  Interventions: Procedure: LAAO

INTERVENTIONS:
Procedure: LAAO — LAAO by use of 3D in silico simulation by FEops HEARTguide as part of the pre-procedural assessment and device size selection

SUMMARY:
The objectives of the current proposal are to analyse to what extend:

1. The use of 3D in silico simulation by FEops HEARTguide improves of influences the pre-procedural assessment and device size selection and to what extend it correlates with final implanted device size and depth compared to TEE, CT and angiography.
2. The use of 3D in silico simulation by FEops HEARTguide increases the operator's confidence in the device size selection.

A total of 100 consecutive patients for the total registry, or 15 to 20 consecutive patients per center, with standard of care follow-up at ±6 weeks and 1 year post procedure.

DETAILED DESCRIPTION:
Left atrial appendage (LAA) occlusion (LAAO) is a well-accepted alternative to oral anticoagulant in the prevention of stroke or systemic thromboembolism in patients with atrial fibrillation (AF).1 While the occlusion is effective, the procedure can sometime be challenging. Part of the challenge is based on the high degree of variability, both at the patient level (anatomy, size, access, filling status etc); and at the device level (different architecture, size, depth, degree of conformity or compression of the device etc.). This is reflected in the percentage change in device sizes of 6.1% to 6.4%; inability to close the LAA 1% to 2.7%; complications such as embolization, tamponade etc.; residual leaks and chances for thrombus formation and subsequent stroke or systemic embolization; lengthy procedures etc.2,3 A well-prepared preprocedural planning addressing the exact anatomy of the left atrial appendage in conjunction with the optimal device size and conformability, results in optimal device selection, reduced instrumentation in the left atrium, faster and safer procedure and optimal final occlusion of the LAA. Different and complimentary techniques are being used by implanting teams, such as transoesophageal echocardiography (TEE), computed tomography (CT) scan, angiography, 3D reconstruction and 3D printing etc.

Some centres are using FEops HEARTguideTM as part of their preprocedural assessment. This is a computational tomography (CT)-based 3D in silico simulation technology suite relying on proprietary computational modelling and simulation techniques, offering physicians detailed preoperative insights into the interaction between transcatheter structural heart devices and the patient's anatomy. It is CE-marked and commercially available on the European and Canadian market. It is currently being used in 81 hospitals in 22 countries.

Belgian Hospitals who are using 3D simulations by FEops HEARTguide as part of their preprocedural assessment are asked to participate to this prospective multicentric registry. The present registry aims to compare all preprocedural imaging tools and to investigate to what extend 3D in silico simulations influences device size selection in LAAO.

The objectives of the current proposal are to analyse to what extend:

1. The use of 3D in silico simulation by FEops HEARTguide improves of influences the pre-procedural assessment and device size selection and to what extend it correlates with final implanted device size and depth compared to TEE, CT and angiography.
2. The use of 3D in silico simulation by FEops HEARTguide increases the operator's confidence in the device size selection.

A total of 100 consecutive patients for the total registry, or 15 to 20 consecutive patients per center, with standard of care follow-up at ±6 weeks and 1 year post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient signed informed consent
* Patient scheduled for LAAO with Amplatzer Amulet (Abbott)
* 3D in silico simulation by FEops HEARTguide available and reviewed before implantation

Exclusion Criteria:

- 3D in silico simulation by FEops HEARTguide not available or not reviewed before implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 consecutive patients, schedule for LAAO with Amplatzer Amulet (Abbott) will be enrolled in this prospective registry after receiving signed informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Improvement in pre-procedural device size selection by use of FEops HEARTguide | At time of procedure
  Correlation between device size selection by use of FEops HEARTguide and implanted device size

CONTACTS AND LOCATIONS:
Overall Officials: Ian Buysschaert, MD, PhD, Principal Investigator — AZ Sint-Jan AV
Locations (6):
- Belgium (6):
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - UZ Brussel, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Maria Middelares, Ghent
  - Sart Tilman - CHU de Liège, Liège

REFERENCES:
- [Derived] De Cock E, Lochy S, Rivero-Ayerza M, Lempereur M, Cornelis K, Debonnaire P, Vermeersch P, Christiaen E, Buysschaert I. Clinical Value of CT-Based 3D Computational Modeling in Left Atrial Appendage Occlusion: An In-Depth Analysis of the PRECISE LAAO Study. Catheter Cardiovasc Interv. 2025 May;105(6):1356-1364. doi: 10.1002/ccd.31464. Epub 2025 Feb 24. PMID 39989438
- [Derived] Swaans MJ, Huijboom MFM, Boersma LVA. Fluoroscopic Guidance: An Echo From the Past? JACC Cardiovasc Interv. 2021 Aug 23;14(16):1827-1829. doi: 10.1016/j.jcin.2021.07.003. No abstract available. PMID 34412800